CLINICAL TRIAL: NCT01691196
Title: Inflammation in Peritoneal Dialysis Patients: Effect of Obesity
Status: Withdrawn | Type: Observational
Why Stopped: Study not initiated
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jerrold S. Levine, Associate Professor of Medicine, University of Illinois at Chicago
Other Study IDs: 2012-0506; Baxter/UIC Ref#2012-04881 (Other: Baxter)
Record Dates: First submitted 2012-09-17; First posted 2012-09-24 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: End-Stage Renal Disease; Renal Disease, End-Stage; Renal Failure, End-Stage; Obesity
Keywords: Obesity; Peritoneal dialysis; Inflammation; Macrophages; Innate immunity
MeSH Terms: conditions — Kidney Failure, Chronic; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Collection: Venous blood after overnight fast will include: (1) heparinized tube (green top) for whole blood (WB) cultures; (2) EDTA tube (lavender top) for CBC and measurement of cytokines and adipokines, and (3) serum-separator (red top) for determination of lipid panel, glucose, insulin, and hemoglobin A1c. Glucose and insulin will be used to calculate HOMA-IR (index of insulin resistance).
  Collection of peritoneal dialysis effluent (PDE): To minimize variability, 2.5% glucose peritoneal dialysis (PD) solution and 4h dwell time will be used for all patients on test day. Immediately after collection, PDE will be chilled before further processing.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our study addresses the following research question: What is the role of obesity in modulating inflammation and innate immune function, as well as the overall responsiveness of innate immune cells (such as macrophages, neutrophils, and other peripheral leukocytes) in patients undergoing peritoneal dialysis?

The investigators hypothesize that obesity will lead to increased inflammation in patients undergoing peritoneal dialysis.

DETAILED DESCRIPTION:
Chronic inflammation is highly prevalent in ESRD and associated with adverse outcomes. For example, chronic exposure of the peritoneal cavity to PD solution leads to induction of cytokines and other inflammatory mediators, generating peritoneal membrane inflammation which results in functional decline of ultrafiltration. Obesity is characterized by a state of chronic low-grade systemic inflammation stemming from expanded adipose tissue mass. Animal studies from our group and others suggest that obesity is associated with exacerbated prolonged inflammatory responses in the peritoneal cavity. The shifting demographic characteristics of the ESRD population, with a rise in elderly patients and those with obesity, is as a significant challenge for management of dialysis patients. Specifically, a 2-fold increase in the percentage of obese patients in the ESRD population has been reported. The caloric burden of PD glucose-containing solutions adds an additional risk for development or exacerbation of obesity and diabetes in patients using this dialysis modality. Few studies have directly evaluated the association between degree of adiposity and inflammation in PD patients. Data obtained from the proposed experiments will help clarify the connection between obesity and risk factors for cardiovascular and infectious diseases in the PD population. These data will also further our knowledge of the basic pathophysiology of both obesity and ESRD and enhance our understanding of factors involved in successful delivery of PD. Results may lead to enhanced nutritional recommendations for PD patients and/or the use of low-glucose or non-glucose alternatives, with a resultant reduction in local and/or systemic inflammation and CVD and other risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years; and
2. peritoneal dialysis (PD) > 6 months.

Exclusion Criteria:

1. infectious episode within 4 weeks; and
2. using immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Plasma and dialysate levels of pro-inflammatory and anti-inflammatory molecules | 24 hours
  Peritoneal dialysate effluent (PDE) and peripheral blood will be obtained from peritoneal dialysis (PD) subjects. Levels of pro- and anti-inflammatory cytokines, chemokines, adipokines, and acute-phase reactants will be evaluated in PDE and plasma. The ability of peripheral leukocytes to respond to microbial stimuli will be studied using whole blood cultures. We predict percentage of body fat will be significantly associated with higher levels of pro-inflammatory factors both systemically and locally and with reduced ability of peripheral leukocytes to respond to microbial stimuli.

SECONDARY OUTCOMES:
Peritoneal macrophage subphenotype | 24 hours
  The composition of leukocytes from peritoneal dialysate effluent (PDE) will be analyzed to evaluate the absolute and relative amounts of leukocyte subclasses. The phenotype of peritoneal macrophages (pMac) will be evaluated by flow cytometry, by real time RT-PCR, and by measurement of mediators characteristic of each activation type following ex vivo culture. We predict that we will observe a significant shift from an anti- to a pro-inflammatory pMac phenotype as adiposity increases

OTHER OUTCOMES:
Measurement of adiposity/obesity | 24 hours
  DXA (dual energy X-ray absorptiometry) will be conducted at UIC body composition laboratory using Hologic 4500 W Elite Scan. Values from DXA scans will be primary method for evaluation of adiposity. Height and weight will be measured by nurse to calculate body mass index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold S Levine, MD, Principal Investigator — UIC; Natalia Litbarg, MD, Principal Investigator — UIC; Giamila Fantuzzi, PhD, Principal Investigator — UIC
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States